CLINICAL TRIAL: NCT05146934
Title: The Relationship Between Hormone Sensitivity and Imaging of Idiopathic Interstitial Pneumonia by Artificial Intelligence
Acronym: IIP
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LM2019173
Record Dates: First submitted 2021-06-30; First posted 2021-12-07 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-06

CONDITIONS: Idiopathic Interstitial Pneumonia
Keywords: Hormone sensitivity; imaging features; artificial intelligence
MeSH Terms: conditions — Idiopathic Interstitial Pneumonias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hormone sensitive group: Prednisone, 0.5mg/kgqd, 3-6months
  Interventions: Radiation: high resolution CT
- Hormone insensitivity group: Prednisone, 0.5mg/kgqd, 3-6months
  Interventions: Radiation: high resolution CT

INTERVENTIONS:
Radiation: high resolution CT — Ground glass，honeycomb，reticulation, consolidation

SUMMARY:
Application of artificial intelligence deep learning algorithm to analyze the relationship between hormone sensitivity of idiopathic interstitial pneumonia and imaging features of high resolution CT.

DETAILED DESCRIPTION:
Methods: the medical records and chest high-resolution CT images of patients with idiopathic interstitial pneumonia admitted to the respiratory department of the Third Hospital of Peking University from June 1, 2012 to December 31, 2020 were retrospectively analyzed.Application of artificial intelligence deep learning neural convolution network method to create recognition technology of different imaging features.Including ground glass, mesh, honeycomb, nodule or consolidation, the model was established. IIP patients were divided into hormone sensitive group and hormone insensitive group according to whether the use of hormone was effective or not.Logistic regression analysis was used to analyze the correlation between statistically significant parameters and hormone sensitivity.Artificial intelligence was used to establish the correlation model between imaging features and clinical data and hormone sensitivity.

ELIGIBILITY:
Inclusion Criteria:

Clinical-pathological-radiology diagnosis of idiopathic interstitial pneumonia Hormone therapy was used; The follow-up data were complete, and the effect of hormone use could be judged.

Exclusion Criteria:

Lung infection disease; Heart failure; Connective tissue disease; IIP Without hormone therapy ; IIP but the follow-up data were incomplete, and the effect of hormone use could not be judged.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From June 1, 2012 to December 31, 2020, all inpatients with IIP were admitted to the respiratory and critical care department of the Third Hospital of Peking University. Total patients are 150, 45 patients using hormone, average age 62 years old, 21 male.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2019-12-30 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
clinical data and imaging feature ratios in both groups | 3-6 months after medication
  clinical data including ages，gender，symptoms,signs,smoking history,complications,laboratory examination，lung function. Imaging feature including ground-glass opacity, reticulation, honeycomb and consolidation.

SECONDARY OUTCOMES:
the relationship between imaging feature ratios and hormone sensibility | 3-6 months after medication
  Logistic regression analyzing the relationship between imaging feature ratios and hormone sensibility.

OTHER OUTCOMES:
development of artificial intelligence algorithm model | 3-6 months after medication
  The U-net method of deep learning convolutional neural network (CNN) was used to create the recognition model of different imaging features. Imaging features include ground-glass opacity, reticulation, honeycomb and consolidation. With the area ratio of imaging features of the two groups as the input and hormone efficacy as the output, the correlation model between imaging features and hormone sensitivity was established by using artificial intelligence k nearest neighbor (KNN) algorithm and support vector machine (SVM) algorithm.

CONTACTS AND LOCATIONS:
Overall Officials: Bei He, Principal Investigator — Peking University Third Hospital Respiratory and critical care department
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No